CLINICAL TRIAL: NCT02604316
Title: SATIN: Satiety Innovation, Study 2. Effect of Novel Fibres (Arabinoxylan and Beta-glucan) in Appetite, Metabolic and Gut Health.
Brief Title: SATIN: Satiety Innovation. Study 2- University of Aberdeen
Acronym: SATIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Københavns Universitet (Other); University of Leeds (Other); University of Liverpool (Other); Universidad de Murcia (Other); University Rovira i Virgili (Other); Karolinska Institutet (Other); Cargill (Industry); The Coca-Cola Company (Industry); Juver Alimentación S.L.U (Industry); Naturex, Spain (Industry); Axxam S.p.A. (Industry); BioActor (Industry); Centro Tecnológico Nacional Agroalimentario Extremadura (Other); Centro Tecnológico Nacional de la Conserva y Alimentación (Other); NIZO Food Research (Other); RTD Services Vienna (Other); ProDigest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2/063/13; 289800 (Other: European Commision); R&D (Other: 2013RW002)
Record Dates: First submitted 2015-03-26; First posted 2015-11-13 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-09

CONDITIONS: Overweight and Obesity
Keywords: Overweight and Obesity; Appetite; Gut hormones and obesity; Arabinoxylan, Beta-Glucan; SmartPill
MeSH Terms: conditions — Overweight; Obesity | interventions — arabinoxylan; beta-Glucans

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arabinoxylan (Experimental): 10 days of weight loss diet calculated as 100% RMR + 15g Arabinoxylan (Medium Chain Naxus, BioActor b.v., Netherlands) per day in incremental dose 25% according energy requirement, 30% protein, 30% fat, 40% carbohydrate
  Interventions: Other: Arabinoxylan
- Control- Non Arabinoxylan (No Intervention): 10 days of weight loss diet calculated 100% RMR using a heterogeneous natural fibre for food ingredients, 30% protein, 30% fat, 40% CHO.
- Beta-Glucan (Experimental): 10 days of weight loss diet calculated as 100% RMR AND 6g Beta-Glucan (Viscofibre, Naturex SA, France) per day in incremental dose 25% according energy requirement, 30% protein, 30% fat, 40%
  Interventions: Other: Beta- Glucan
- Control Non Beta glucan (No Intervention): 10 days of weight loss diet calculated 100% RMR using a heterogeneous natural fibre for food ingredients, 30% protein, 30% fat, 40% CHO.

INTERVENTIONS:
Other: Arabinoxylan — 10 days of weight loss diet calculated as 100% RMR + 15g Arabinoxylan (Medium Chain Naxus, BioActor b.v., Netherlands) per day in incremental dose 25% according energy requirement, 30% protein, 30% fat, 40% carbohydrate.
  Other Names: MC- NAXUS
  Arms: Arabinoxylan
Other: Beta- Glucan — 10 days of weight loss diet calculated as 100% RMR + 6g β-glucan (Viscofibre, Naturex SA, France) per day in incremental dose 25% according energy requirement, 30% protein, 30% fat, 40%
  Other Names: Viscofiber
  Arms: Beta-Glucan

SUMMARY:
The proposed study will address the effect of developed novel food products through processing innovation on motivation to eat, biomarkers of satiety, nutrient bioavailability and gut health using in vivo studies and validating new in vivo approaches.

Specifically in this protocol the investigators will address, in a short human intervention study the effect of a potentially satiating product on appetite, appetite biomarkers, particularly the influence on gut microbiota, tolerance and safety of the products in healthy obese and overweight participants in free living conditions.

DETAILED DESCRIPTION:
Previous research has suggested that food structure and food composition has a role to play in controlling consumption. Low-energy, high-fibre diets provide physical bulk in the gastro-intestinal tract to sustain fullness in a way that low-volume, energy-dense foods cannot. However, studies shown low long term acceptability be probably associated to its poor palatability. Taste and hedonic experience remain the main drivers of consumer choice, and the immediate sensory aspect of food products such as palatability to have greater salience to consumers than their health promoting properties.

Changing the properties of foods merely by changing oro-sensory properties and through the delay of gastric emptying deals with mechanisms critical to within-meal satiation and early post meal satiety and may produce only transient suppression of hunger unless regularly consumed and represent benefits in delivering nutritional stimuli to key parts of the gastro-intestinal tract. The potential to manufacture change can make food structure variety now seem near limitless due the numerous advances in food technology.

Several recent reports have associated satiety effects with fermentable fibre sources in human dietary studies. Apparently, the large intestine microbiota recovers 'extra' calories from the diet and might contributes to obesity. However, the different mechanisms involved in lean and obese subjects are not completely resolved. Recent evidence in experimental animal designs indicates that changes in gut microbiota composition may be associated with increased food intake and obesity suggesting that satiety and intake are influenced by the species composition of the gut microbiota.

This short-term human nutrition study comprises in a randomised, cross-over design testing either two potentially satiety product, Arabinoxylan (A) or Beta-glucan (B) against an equivalent amount of heterogeneous natural fibre (Control) in 40 healthy-obese volunteers, aged 18-65 years old, BMI between 27 and 42Kg/m2 from both genders after an initial maintenance diet in free- living conditions.

Dietary intake, body weight, blood pressure would be monitored through the study. Faecal, urine and blood samples will be collected to monitor, glucose, insulin, gut peptides and assess metabolites of dietary and microbial origin. Orocecal Transit Time (OCTT), carbohydrate fermentability and methanogen status will be estimated using a breath test and transit time will be determined using SmartPill™.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18-65 years old
* Body Mass Index (BMI) 27-42kg/m2
* Overall healthy
* Weight Stable (<3 kg change in the past 4 months, before the trial).

Exclusion Criteria:

* Medical:
* Heavy smokers (more than 10 cigarettes/day) or heavy alcohol consumers (more than 4 alcohol units/day for male and more than 3 alcohol units/day for female).
* Obesity of endocrine origin.
* Chronic metabolic conditions: diabetes, hepatic disease, gout, kidney, thyroid or coagulation disease.
* Gastrointestinal disorders: celiac disease, Intenstinal Bowel Disease (IBD), irritable bowel syndrome (IBS), chronic constipation, diverticulitis, history of gastric bezoar. Suspected strictures, fistulas, or physiological GI obstruction.
* Psychiatric disorder: severe depression, bulimia, anorexia, schizophrenia, bipolar disorder.
* Gastrointestinal procedure or surgery in the past three months.
* Disorders of swallowing, severe dysphagia to food or pills.
* Pregnancy

Medication exclusion criteria

* Appetite modulator drugs: orlistat, sibutramine, rimonabant.
* Mood disorder medications: antidepressants, lithium.
* Others: oral antidiabetics, insulin, digoxin, thyroid hormones, antibiotics, steroids or immunosuppressants, recreational substances.
* Use of implanted or portable electro-mechanical device such as cardiac peacemaker or infusion pump.
* Blood donor in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Effect of Arabinoxylan or Beta- Glucan on weight loss and body composition | 72 hours
  During this part of the study the effect of novel fibre of 3 dietary interventions subsequent each other: Maintenance (3 days), Arabinoxylan or Beta glucan per 10 days and Control diet per 10 days. Weight loss will be assessed after dietary intervention. Changes on body weight, BMI and total and regional body composition information using a two compartment model (fat mass and fat free mass by air displacement densitometry -Bod-Pod) will be assessed at the end of each dietary intervention. Resting Metabolic Rate will be assessed the beginning and at the end of the weight loss diet (Deltatrac).

SECONDARY OUTCOMES:
Effect of Arabinoxylan or Beta- Glucan on gut health | 23 days
  The effect of a novel fibre on gut health: Gut microbiota, short chain fatty acids production.
  To assess metabolites of dietary and microbial origin including short chain fatty acid. Bacterial community structure will be assessed by targeted quantitative polymerase chain reaction (qPCR), high throughput 454 sequencing (Walker et al., ISME J 2010) and 4',6-diamidino-2-phenylindole (DAPI) staining to estimate total bacteria. Gut transit will be assessed once at the end of each diet using a wireless motility device (SmartPill™). Only 4 volunteers will receive this assessment during the last 5 days of each maintenance period.
  Questionnaires will be provided to monitor qualitatively gastrointestinal wellbeing during each dietary intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Alexandra M Johnstone, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Rowett Institute of Nutrition and Health. University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- See also: SATIN-EU Consortium web page — http://www.satin-satiety.eu/